CLINICAL TRIAL: NCT07283770
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Dose Escalation Study Evaluating Safety and Pharmacokinetics of VX-581 in Healthy Subjects
Brief Title: Dose Escalation Study Evaluating the Safety and Pharmacokinetics of VX-581 in Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX25-581-001
Record Dates: First submitted 2025-12-04; First posted 2025-12-16 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A: Single Ascending Dose (Experimental): Participants will be randomized to receive a single dose of VX-581.
  Interventions: Drug: VX-581
- Placebo: Part A (Placebo Comparator): Participants will be randomized to receive a single dose of placebo matched to VX-581.
  Interventions: Drug: Placebo
- Part B: Multiple Ascending Dose (Experimental): Participants will be randomized to receive multiple doses of VX-581.
  Interventions: Drug: VX-581
- Placebo: Part B (Placebo Comparator): Participants will be randomized to receive multiple doses of placebo matched to VX-581.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VX-581 — Suspension for Oral Administration.
  Arms: Part A: Single Ascending Dose; Part B: Multiple Ascending Dose
Drug: Placebo — Suspension for Oral Administration.
  Arms: Placebo: Part A; Placebo: Part B

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics of single and multiple ascending doses of VX-581.

DETAILED DESCRIPTION:
The study is being conducted to evaluate the safety, tolerability, and pharmacokinetics of single and multiple ascending doses of VX-581 in healthy participants and consists of Screening Phase, Treatment Phase and Safety Follow-up Phase. Note: This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index (BMI) of 18.0 to 32.0 kilogram per meter square (kg/m^2)
* A total body weight of more than (>) 50 kg
* Male and Female participants of non-childbearing potential

Key Exclusion Criteria:

* History of febrile illness or other acute illness that has not fully resolved within 14 days before the first dose of study drug
* Any condition possibly affecting drug absorption

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-12-09 (Actual); Primary Completion 2026-11-19 (Estimated); Study Completion 2026-11-19 (Estimated)

PRIMARY OUTCOMES:
Part A: Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day -1 up to Day 34
Part B: Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day -1 up to Day 66

SECONDARY OUTCOMES:
Part A: Maximum Observed Plasma Concentration (Cmax) of VX-581 | From Day 1 up to Day 34
Part A: Area Under the Concentration Versus Time Curve From the Time of Dosing Up to 24 Hours (AUC0-24h) of VX-581 | From Day 1 up to Day 34
Part B: Maximum Observed Plasma Concentration (Cmax) of VX-581 | From Day 1 up to Day 66
Part B: Area Under the Concentration Versus Time Curve From the Time of Dosing Up to 24 Hours (AUC0-24h) of VX-581 | From Day 1 up to Day 66

CONTACTS AND LOCATIONS:
Locations (1):
- Altasciences - Kansas City, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/our-science/clinical-trials-data-sharing/